CLINICAL TRIAL: NCT05391425
Title: The Effect of Solifenacin Used for Lower Urinary Tract Symptoms on Sexual Function in Premenopausal vs Postmenopausal Women: A Prospective Observational Study
Brief Title: The Effect of Solifenacin Used for Lower Urinary Tract Symptoms on Sexual Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Collaborators: Arnavutkoy State Hospital (Other)
Responsible Party: Principal Investigator, inci sema tas, MD, Istanbul University
Other Study IDs: solifenacinpm
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Urge Incontinence; Urgency-frequency Syndrome
Keywords: urgency; urge urinary incontinence; solifenacin; sexual function; menopause; anticholinergic
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- premenopausal: Premenopausal patients, presented in Arnavutkoy State Hospital Gynecology Clinic with lower urinary tract symptoms that will be treated with Solifenacin (Vesicare 5mg).
  Interventions: Other: no intervention
- postmenopausal: Postmenopausal patients, presented in Arnavutkoy State Hospital Gynecology Clinic with lower urinary tract symptoms that will be treated with Solifenacin (Vesicare 5mg).
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention planned, since it is an observational study

SUMMARY:
This study aims to determine whether Solifenacine used for lower urinary tract symptoms improves sexual function and if so does this improvement differs between premenopausal and postmenopausal women.

DETAILED DESCRIPTION:
Solifenacin is an anticholinergic drug that is commonly used for lower urinary tract symptoms such as urgency, frequency and urge urinary incontinence. Solifenacin use and sexual function improvement is presented in some research, but the correlation between the improvement in sexual function and LUTS symptoms is yet not investigated. Also the effect on sexual function in premenopausal vs postmenopausal women are unknown.

ELIGIBILITY:
Inclusion Criteria:

* Women presented in Arnavutkoy State Hospital Gynecology Clinic with lower urinary tract symptoms that are planned to start treatment with Solifenacin 5 mg (Vesicare 5mg).
* Patients agreed to involve in the study, having discussed other treatment options and possible side effects of the medication.
* Informed consent obtained

Exclusion Criteria:

* urinary tract infection
* stress urinary incontinence
* urinary retention
* grade 2 or above pelvic organ prolapse according to POP-Q scale
* Solifenacin contraindications such as narrow angle glaucoma, allergy of Solifenacin or other components of the drug.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women presented in Arnavutkoy State Hospital Gynecology Clinic with lower urinary tract symptoms that are planned to start treatment with Solifenacin 5 mg (Vesicare 5mg) are enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-06-03 (Estimated); Study Completion 2024-06-03 (Estimated)

PRIMARY OUTCOMES:
the effect of solifenasin used for lower urinary tract symptoms on sexual function | 6 months
  Female Sexual Function Index (FSFI) scores change between in baseline, 3 and 6 months after Solifenacin use for lower urinary tract symptoms.
the effect of solifenasin used for lower urinary tract symptoms on sexual function in premenapausal vs postmenapausal women | 6 months
  The aim of this study is to determine whether Solifenacine used for lower urinary tract symptoms improve sexual function (measured by Female Sexual Function Index; higher scores meaning sexual dysfunction with the cut off value of 26.) and if so does this improvement differs between premenaupausal and postmenaupausal women.

SECONDARY OUTCOMES:
the effect of Solifenacin treatment for lower urinary tract symptoms (LUTS) on sexual function and its correleation with the improvement in LUTS | 3 and 6 months
  The aim of this study is to determine whether Solifenacine used for lower urinary tract symptoms improve sexual function (measured by Female Sexual Function Index; higher scores meaning sexual dysfunction with the cut off value 26.)and if so does this correlates with the improvement with lower urinary tract disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Arnavutkoy State Hospital, Istanbul, Arnavutkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided